CLINICAL TRIAL: NCT00466908
Title: Accuracy of the Pentacam and IOL Master to Calculate the Effective Corneal Power After Corneal Refractive Surgery
Status: Withdrawn | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Kerry S. Solomon, Medcial University of South Carolina
Other Study IDs: MRC-07-001
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2010-10

CONDITIONS: Cataract Extraction; Refractive Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pentacam and IOL Master — Pentacam and IOL Master

SUMMARY:
The purpose of this study is to determine the accuracy of the Pentacam and IOL Master to calculate the effective corneal power (keratometry, corneal curvature) in patients who have undergone both corneal refractive surgery and lens extraction with intraocular lens implantation.

DETAILED DESCRIPTION:
The accuracy of IOL calculation is important for the visual outcome of patients undergoing cataract extraction and IOL implantation. Different formulas such as Holladay I, HofferQ, SRKT have been used with excellent results. All formulas use the corneal power among other factors to calculate the IOL power. Corneal refractive surgery i.e. radial keratotomy (RK), photorefractive keratectomy (PRK), and Laser in situ keratomileusis (LASIK) changes the corneal power; therefore, it is difficult to measure the true corneal power after surgery by any form of direct measurement, such as keratometry, or corneal topography. Keratometry and topography assume a normal relationship between the anterior and posterior corneal curvatures, and measure the anterior corneal radius. RK for myopia flattens both the anterior corneal radius and the posterior corneal radius while PRK and LASIK for myopia flattens the anterior corneal radius but leaves the posterior corneal radius mostly unchanged.

Standard keratometry measures an intermediate area and extrapolates the central power based on some very broad assumptions. For this reason, keratometry, autokeratometry and simulated keratometry by topography will typically over-estimate central corneal power following keratorefractive surgery for myopia. This inaccuracy leads to an inability to meet the patients' rising expectations and with the increasing popularity of refractive surgery, calculating intraocular lens (IOL) power after refractive surgery is becoming increasingly important.

Different methods to calculate the effective corneal power (keratometry) after refractive surgery have been described (historical data, effective refractive power, modified Maloney method, etc), however, intraocular lens power calculations in eyes with previous refractive surgery remains difficult because of the inaccuracy of keratometry power measurements.

The Pentacam (Comprehensive Eye Scanner) is a non-invasive, diagnostic system created to take photographs of the anterior segment of the eye by a rotating Scheimpflug camera measurement. This rotating process supplies pictures in three dimensions. The center of the cornea is measured very precisely because of this rotational imaging process. The measurement process lasts less than two seconds and minute eye movements are captured and corrected simultaneously. By measuring 25,000 true elevation points, precise representation, repeatability and analysis are guaranteed. It provides a topographic analysis of the corneal front and back surfaces that is based on the true elevation measurement from limbus to limbus. Both corneal surfaces can be selected for analysis in axial (sagittal), tangential or elevation representation modes.

The Pentacam using tomography calculates a virtual model of the anterior segment of the eye. It is possible to move, zoom and rotate it to detect e.g. iris defects, cornea incisions e.g. RK or size, location and shape of opacifications in the crystalline lens. The slicing function in the three dimensions offers a detailed view of the different layers of the eye. It includes the Holladay report that was developed to improve the calculation of IOLs for patients which have undergone corneal refractive surgery.

The IOL Master is a non-contact optical coherence biometry that makes possible the exact measurement of visual axis length. Its accuracy is not affected by high ametropia, pupil size or state of accommodation. This non-contact technology makes it easy on the patient: no local anesthesia, water bath, or contact probe. For IOL power calculation after previous refractive corneal surgery, one can derive the effective corneal power using either the clinical history method, or the rigid contact lens over-refraction method. It therefore permits selection of a suitable lens after myopic LASIK/PRK without requiring refractive pre-LASIK data or additional contact lens over-refraction.

The purpose of this study is to determine the accuracy of the Pentacam and IOL Master to calculate the effective corneal power (keratometry, corneal curvature) in patients who have undergone both corneal refractive surgery and lens extraction with intraocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have undergone corneal refractive surgery (RK, PRK or LASIK) prior to cataract extraction.
* Age: 40 to 80 years old.
* Subjects must have undergone cataract extraction at least 4 weeks prior to enrollment in this trial.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphtalmus or macrophtalmus, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery (other than cataract extraction) within the past three months or intraocular laser surgery within one month in the operated eye.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject must have undergone corneal refractive surgery (RK, PRK or LASIK) prior to cataract extraction.
  Age: 40 to 80 years old.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helga Sandoval, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina, United States